CLINICAL TRIAL: NCT06975423
Title: Somatosensory Feedback to Improve Neural Control of Walking in Older Adults
Brief Title: Walking Sensation Study
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: The Claude D. Pepper Older Americans Independence Centers (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Treatment
Other Study IDs: IRB202500632; 5P30AG028740 (NIH)
Record Dates: First submitted 2025-05-07; First posted 2025-05-16 (Actual); Last update posted 2026-02-09 (Actual); Status verified 2025-09

CONDITIONS: Aging; Sensory Deficit
Keywords: Dual-task walking; Brain activity; Walking performance

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes | Unapproved Device: Yes | US Export: Yes

ARMS (2):
- Active lower-limb neuroprosthesis (Active Comparator): Participants will perform single- and dual-task walking trials, including Serial 7 Subtraction, with and without navigating wide and high obstacles (to increase cognitive effort), while wearing Walkasins in "ON" setting
  Interventions: Device: Active lower-limb neuroprosthesis
- Inactive lower-limb neuroprosthesis (Sham Comparator): Participants will perform single- and dual-task walking trials, including Serial 7 Subtraction, with and without navigating wide and high obstacles (to increase cognitive effort), while wearing Walkasins in "OFF" setting
  Interventions: Device: Inactive lower-limb neuroprosthesis

INTERVENTIONS:
Device: Active lower-limb neuroprosthesis — Walkasins sensory neuroprosthesis provides real-time sensory input by delivering vibrotactile stimuli to the lower limbs above the ankle
  Arms: Active lower-limb neuroprosthesis
Device: Inactive lower-limb neuroprosthesis — Walkasins sensory neuroprosthesis does not provide real-time sensory input by delivering vibrotactile stimuli to the lower limbs above the ankle
  Arms: Inactive lower-limb neuroprosthesis

SUMMARY:
The primary objective of this new line of research is to test whether augmenting sensory information from the legs, using Walkasins sensory neuroprosthesis, can enhance performance of a complex walking task in older adults with foot sensory impairment. The overarching hypothesis is that Walkasins will enhance the automaticity and reduce cognitive demand of walking in older adults with foot sensory impairments, as measured by reduced prefrontal activity, decreased dual-task costs, and lower gait variability.

DETAILED DESCRIPTION:
Preserving mobility function in older adults is crucial for ensuring safe walking in complex environments, including home and community settings. A common example is navigating a busy street with obstacles like uneven sidewalks and pedestrians, or a home with furniture, stairs, and narrow hallways, all while engaging in a conversation or mental task. Such environments create a potential risk for older adults, who may show declines in function across multiple systems, including sensation, cognition, and mobility. Successfully walking in complex environments depends on cognitive control processes, such as attention and motor planning, which rely on sufficient sensory information from peripheral receptors. Somatosensory impairment, particularly in the feet, is common among older adults and tends to increase progressively with age, often worsened by the presence of certain diseases. Age-related somatosensory impairments disrupt essential input to central motor and cognitive networks, raising the risk of accidental collisions, slips, trips, and injurious falls. Older adults may compensate by increasing cognitive load (attention and executive control of movement). However, this shift may overburden cognitive systems, again raising the risk of collisions, slips, trips, and falls. There is a critical, yet underexplored, need to restore somatosensory input to the nervous system during walking in older adults with foot sensory impairments. Therefore, the objective of this study is to investigate whether the use of a novel lower-limb sensory prosthesis, Walkasins, improves complex walking performance and reduces cognitive load. This crossover study will enroll 30 participants with foot sensory impairment, who will undergo complex walking performance assessments while wearing the Walkasins in both the "on" and "off" settings. These settings will be assessed in separate visits occurring at least one week apart, to allow for a washout period. The walking course will use a pressure-sensitive instrumented walkway to analyze kinetic and kinematic variability of the gait pattern. These assessments will include typical walking, as well as dual-task walking with and without obstacle crossing as a behavioral assessment of cognitive load. Furthermore, cognitive load will be assessed by measuring prefrontal cortical activity with functional near infrared spectroscopy (fNIRS). We will address the following specific aims:

Specific Aim 1 is to test whether Walkasins can improve walking performance, hypothesizing greater reductions in dual-task costs and gait variability when using Walkasins in the "on" setting compared to the "off" setting.

Specific Aim 2 is to assess the potential of Walkasins to reduce cognitive load during walking, hypothesizing lower prefrontal cortical activity when using Walkasins in the "on" setting compared to the "off" setting.

This pilot study enhances our understanding of age-related sensory impairments in neural control and walking performance and will prepare us for larger-scale trials with more intervention sessions, larger sample sizes, and a focus on the underlying neurophysiological mechanisms. This study and future research contribute to the development of rehabilitation strategies that support healthy aging and enhance functional mobility.

ELIGIBILITY:
Inclusion Criteria:

* Not having any significant existing medical conditions, historical health issues, or medications (outlined in the exclusion criteria table above) that could impede the execution of the walking task and assessment.
* age 65 - 95.
* no severe high blood pressure (systolic < 180 mmHg and/or diastolic < 100 mmHg at rest).
* no severe vision impairment: visual acuity ≥ 20/70 as determined by Snellen eye chart.
* slow walking speed: preferred walking speed slower than 1.0 m/s over 10 meter.
* no cognitive impairment: Montreal Cognitive Assessment (MoCA) score ≥ 26 out of 30 possible points.
* foot sensory impairment: Inability to feel the 10 g monofilament at ≥1 of 10 tested sites on either foot is considered a sign of impaired protective sensation. loss.

Exclusion Criteria:

* diagnosed neurological disorder or injury of the central nervous system, or observation of symptoms consistent with such a condition (Alzheimer's, Parkinson's, stroke, etc.)
* severe arthritis, such as awaiting joint replacement
* current cardiovascular, lung or renal disease; untreated diabetes; terminal illness
* myocardial infarction or major heart surgery in the previous year
* cancer treatment in the past year, except for nonmelanoma skin cancers and cancers having an excellent prognosis (e.g., early stage breast or prostate cancer)
* current diagnosis of schizophrenia, other psychotic disorders, or bipolar disorder
* currently taking medications that affect the central nervous system, such as benzodiazepines, anti-cholinergic medication, and GABAergic medication, among others
* no severe vision impairment (visual acuity ≥ 20/70 as determined by Snellen eye chart)
* uncontrolled hypertension at rest (systolic > 180 mmHg and/or diastolic > 100 mmHg)
* bone fracture or joint replacement in the previous six months
* current enrollment in any other clinical trial
* planning to relocate out of the area during the study period
* non-English* speaking, due to the likelihood of difficulties following instructions and communicating remotely
* clinical judgment of the investigative team

Ages: 65 Years to 95 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Older Adult
Enrollment: 30 (Estimated)
Dates: Start 2025-09-08 (Actual); Primary Completion 2027-01-31 (Estimated); Study Completion 2027-03-31 (Estimated)

PRIMARY OUTCOMES:
Dual-Task Cost | Baseline, 7-day follow-up
  Comparison of dual-task walking performance between active and inactive lower-limb neuroprosthesis conditions
Gait Variability | Baseline, 7-day follow-up
  Comparison of gait performance between active and inactive lower-limb neuroprosthesis conditions.
Brain Activity | Baseline, 7-day follow-up
  Comparison of prefrontal cortical activity during active versus inactive lower-limb neuroprosthesis conditions.

SECONDARY OUTCOMES:
Kinematic and Dynamic Movement | Baseline, 7-day follow-up
  Comparison of kinematic and dynamic movement during active versus inactive lower-limb neuroprosthesis conditions.

CONTACTS AND LOCATIONS:
Locations (1):
- Clinical and Translational Research Building, Gainesville, Florida, United States

IPD SHARING:
Plan to Share IPD: Yes
Supporting Information: Study Protocol, CSR